CLINICAL TRIAL: NCT02157090
Title: Clinical Assessment of the Effectiveness and Safety of Herpes Patch SOS (Hansaplast®) Based on Hydrocolloids Without Active Substances in the Treatment of Herpes Simplex Labialis in Comparison to a Competitor's Product (Herpes Vesicle Patch of COMPEED®)
Brief Title: Clinical Assessment of the Effectiveness and Safety of Herpes Patch SOS in the Treatment of Herpes Simplex Labialis in Comparison to a Competitor's Product.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Beiersdorf AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: Herpes patch study 32583
Record Dates: First submitted 2010-10-28; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Herpes Simplex Labialis
Keywords: HSL of lips; perioral skin; duration of HSL symptoms not more than three days; not acyclovir or other cold sore therapies
MeSH Terms: conditions — Herpes Labialis

ARMS (2):
- Herpes Patch SOS (Hansaplast®) (Active Comparator)
  Interventions: Other: Herpes Patch SOS (Hansaplast®)
- Herpes vesicle patch of Compeed® (Active Comparator)
  Interventions: Other: Herpes vesicle patch of Compeed®

INTERVENTIONS:
Other: Herpes Patch SOS (Hansaplast®)
  Arms: Herpes Patch SOS (Hansaplast®)
Other: Herpes vesicle patch of Compeed®
  Arms: Herpes vesicle patch of Compeed®

SUMMARY:
Recent clinical studies showed, that a hydrocolloid patch is effective, well tolerated and comparable with aciclovir cream 5 % for the treatment of HSL lesions, while affording additional benefits of wound protection, discretion and relief of social embarrassment. The aim of the actual study was the clinical assessment of the effectiveness and safety of Hansaplast® SOS Herpes Patch (HPHP) in comparison to Compeed® Herpes Vesicle Patch (CHP) in treating HSL. Both products are CE-certificated and are available at the market for medical devices.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* with a history of recurrent HSL of the lips and/or perioral skin
* lesions typically manifesting as classical lesions
* duration of HSL symptoms not more than three days
* haven´t used acyclovir or other cold sore therapies

Exclusion Criteria:

* pregnancy
* lactating women
* women of child-bearing age without medically secured contraceptions
* topical or systemic therapy with analgesic
* anti-inflammatory or antiviral agents within the last 2 weeks
* topical therapy within the treatment area
* systemic therapy with cytostatics or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study was the Subjects Global Assessment of Therapy (SGAT) at final visit.

SECONDARY OUTCOMES:
Number of patients with healed HSL lesions on day 5 and day 10 (assessed by clinician)
Blinded clinician global assessment (IGAT) at the end of therapy.
Development of lesion size.
The number of study subjects with vesicles at onset of the study and at visit 2 and the final visit 3.
Clinician-assessed lesion stage at onset of the study and at visit 2 and the final visit 3.
Clinician-assessed time to complete healing from begin of the study.
Time to complete healing of HSL after beginning of signs and symptoms.
Assessment of the local compatibility by patient and by investigator.
The severity and duration of subject-assessed individual signs and symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Carl Gustav Carus at the Technische Universität Dresden, Dresden, Saxony, Germany